CLINICAL TRIAL: NCT06431984
Title: Kit de Pharmacologie Spatial - Analyse de l'Utilisation Des Dried Blood Spot Pour le Dosage de la caféine Chez Des Volontaires Sains en microgravité au Cours Des Vols Paraboliques
Brief Title: Pharmacology Space Kit (PSK) - Dried Blood Spot for Caffeine Pharmacokinetics Under Microgravity Conditions
Acronym: PSK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C22-80; 2022-A02794-39 (Registry Identifier: IDRCB)
Record Dates: First submitted 2024-05-15; First posted 2024-05-29 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2024-05

CONDITIONS: Drug Mechanism; Metabolism Medication Toxicity; Space Motion Sickness
MeSH Terms: conditions — Space Motion Sickness | interventions — Patch Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healthy subjects (Experimental): Participants are healthy volunteers selected by the investigating team. The size of the study is limited by the number of individuals authorised to board the aircraft.
  The flying participants in the experiment will be the aircraft crew, i.e. volunteers from the research teams taking part in the parabolic flight.
  Healthy volunteers over the age of majority will be included in the study.
  Interventions: Diagnostic Test: prick test

INTERVENTIONS:
Diagnostic Test: prick test — self-sampling of capillary blood using the finger prick test method

SUMMARY:
The PSK study is preliminary to the study of drug metabolism in space flight conditions. The investigators propose to use simplified blood sampling methods that can be applied in microgravity. This method is based on the use of capillary blood, obtained using an automatic lancet for diabetics, the blood droplet then being deposited on specific blotting paper, and then studied in the laboratory. In 2022, the investigators validated the transfer of artificial blood in parabolic flight conditions, as well as the validity of cardiovascular drug dosage.

The objective of the 2023 study is to validate the collection and transfer of capillary blood, on themselves, by healthy volunteers with little training, for the blood dosage of caffeine after intake of standard doses of alimentary caffeine.

The primary objective is a feasibility of 90% of sampling in microgravity, compared with 95% on ground. Secondary objectives are the pharmacokinetic of different forms of caffeine, according to genetic background and other modifiers of CYP1A2.

DETAILED DESCRIPTION:
The investigators propose to use simplified blood sampling methods that can be applied in microgravity. This method is based on the use of capillary blood, obtained using an automatic lancet for diabetics, the blood droplet then being deposited on specific blotting paper, and then studied in the laboratory.

The objective of the study is to validate the collection and transfer of capillary blood from finger prick test, performed on themselves, by healthy volunteers after a short training, for the blood dosage of caffeine. Dietary caffeine will be used, issued from standardized espresso, tea or dark chocolate.

Caffeine is a universally used food substance and is metabolised by a pathway common to many drugs (CYP 1A2). The aim is to show that it is possible to collect blood in this way, and to carry out assays of caffeine. Secondary objectives are to assess the kinetics of caffeine metabolism through the metabolic ratio (AUC paraxanthine/AUC caffeine), and to correlate these kinetics with genetic variations in CYP 1A2 activity.

Participants are healthy volunteers already selected to take part in the parabolic flight campaign.

A success rate of 95% for ground sampling, and 90% for in-flight sampling is assumed as satisfactory. If 5 volunteer participants during the 3 days of flying carry out 2 in-flight samplings, this results in 30 in-flight samplings. If the other 25 flying volunteers take only one in-flight sample, means 25 in-flight samples (total 55). On the ground, the 30 volunteers will take 90 samples, for a total of 145 minimum samples. An equivalence threshold for a maximum 20% difference between flight and ground conditions is considered. For a difference of 10, 15 and 20%, the power is 34, 79 and 97% respectively. It can therefore conclude that the difference between the two sampling conditions is not clinically significant.

ELIGIBILITY:
Inclusion Criteria:

* Be affiliated to a social security scheme or benefit from such a scheme.
* Have obtained a medical certificate stating that they are fit for parabolic flights.
* Be aged between 18 and 70
* Be in good health: no chronic treatment that could interact with the metabolism of caffeine, no progressive disease
* Must not have any contraindications to taking caffeine (30 to 100 mg). Volunteers will also be asked not to consume caffeine (coffee, chocolate, energy drinks, tea, cola, etc.) in the 24 hours preceding the experiment.

Exclusion Criteria:

* Be the subject of a legal protection measure (safeguard of justice, curatorship or guardianship)
* suffer from haematophobia (irrational fear of blood)
* Have a current infectious disease, particularly viral
* Have an active chronic illness
* Have a high usual intake of caffeine (>4 espressos, >4 cups of tea, >100g dark chocolate per day)
* Total intolerance to all forms of caffeine
* Smoke more than 20 cigarettes a day
* Have weaned themselves off smoking for less than a month
* Have a history of severe Raynaud's phenomenon
* Have a history of naupathy
* Suffering from naupathy during a flight

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
Percentage of valid capillary blood deposit on dry support | through study completion, an average of 3 days
  A blood transfer is considered as successful IF the 3 following criteria are fulfilled
  1. Blood spot covering > 8 mm2 (3 mm punch circle)
  2. Obtaining a drop of blood within the allotted time of 22 sec of microgravity
  3. The drop is neither smeared nor smashed on the blotting paper

SECONDARY OUTCOMES:
Identification of factors leading to self-sampling failure a. Time too short b. Insufficient drop c. Inadequate transfer | through study completion, an average of 1 year
  Identification of self-sampling failure factors
  * Deposition time in flight > 22 seconds of weightlessness
  * Blood stain covering 80% or more of the reference circle: diameter of the stain taken by photography
Caffeine kinetic under different formulations and dosages | through study completion, an average of 3 days
  Area under the curve of caffeine and paraxanthine, metabolic ratio (para/caffeine)
Caffeine kinetic under different CYP1A2 genotypes | through study completion, an average of 3 days
  Area under the curve of caffeine and paraxanthine, metabolic ratio (para/caffeine)
Caffeine kinetic under different gravity conditions | through study completion, an average of 3 days
  Area under the curve of caffeine and paraxanthine, metabolic ratio (para/caffeine)
Acceptability | through study completion, an average of 1 year
  A paper questionnaire will be handed out just after the parabolic flight at the time of the last sampling. It will be made up of closed questions based on 3 dimensions of satisfaction:
  * The quality of the information given by the investigating team on the capillary blood sampling process in order to improve our paper-based operating procedure.
  * Their physical and psychological well-being during the finger prick test demonstration phase before the flight, during the flight and at the end of the flight campaign to ensure that the participants felt comfortable and confident in the sampling situation.
  * Assessment of their performance during the study in flight and on the ground, and whether they would be interested in self-sampling for a future space mission.
Stability of dry blood spots | through study completion, an average of 1 year
  Area under the curve of caffeine and paraxanthin, metabolic ratio (para/caffeine) at 6 months interval
  * Visual appearance (degradation, colour change, etc.)
  * Comparison of relative areas obtained during the study with those obtained in a conventional laboratory situation

CONTACTS AND LOCATIONS:
Locations (1):
- AIRBUS A 310 - Zero-G, Mérignac, France

REFERENCES:
- [Background] Derobertmasure A, Toh LS, Verstuyft C, Lukic S, De Sousa Carvalho C, Couronne R, Beauvalet M, Chhun S, Boutouyrie P. Feasibility of dried blood spot collection for caffeine pharmacokinetic studies in microgravity: Insights from parabolic flight campaigns. Br J Clin Pharmacol. 2026 Jan;92(1):35-47. doi: 10.1111/bcp.16320. Epub 2024 Oct 29. PMID 39473131